CLINICAL TRIAL: NCT03607578
Title: Test of Developed Interventions to Prevent Skin Cancer: a Randomized Study Targeting Danes Going on Vacation to Sunny Destinations With High UV Index
Brief Title: Test of Interventions to Prevent Skin Cancer Among Danes on Vacation in High UV Index Sunny Destinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Køster (Other)
Responsible Party: Sponsor-Investigator, Brian Køster, Research scientist, Danish Cancer Society
Organization: Danish Cancer Society (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RCT429-2015-294
Record Dates: First submitted 2018-02-20; First posted 2018-07-31 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Sunburn; Ultraviolet Radiation Exposure; Skin Cancer; Malignant Melanoma; Non-melanoma Skin Cancer; Keratinocyte Skin Cancer
Keywords: Prevention
MeSH Terms: conditions — Sunburn; Skin Neoplasms; Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group - Minimal Intervention (Other): Minimal intervention
  Interventions: Behavioral: Other: Control Group - Minimal Intervention
- Protection Routine 1 (Experimental)
  Interventions: Behavioral: Experimental: Protection Routine 1
- Protection Routine 2 (Experimental)
  Interventions: Behavioral: Experimental: Protection Routine 2
- Protection Routine 1+2 (Experimental)
  Interventions: Behavioral: Experimental: Protection Routine 1; Behavioral: Experimental: Protection Routine 2

INTERVENTIONS:
Behavioral: Other: Control Group - Minimal Intervention — Basic Campaign Folder
  Arms: Control Group - Minimal Intervention
Behavioral: Experimental: Protection Routine 1 — New folder, sun advice of Danish Sun Safety Campaign, rationale, prioritization, overview of sun prevention. Activity planner with outdoor activities like bathing, sports and excursions before and after noon (UVI maximum) and indoor activities; shopping, lunch, relaxation and transportation in middle of day and possibility to plan vacation to minimize risk. Instructions for download of UV-App includes use of alert, and information about the features of the app; how to be informed of current UV risk before and during vacation. Link for download of the app is sent by text-message and e-mail. Skintype guide is included in the app and as an individual entity. It includes scoring questions about tan and burn reaction in the sun, a color scale, eye and hair color and freckles. Participants get a description of their skin type and examples of time their particular skin type will resist the sun before erythema occurs at particular UV-levels and functions as an eye-opener.
  Other Names: Intensive information and training in current advice - UVI & Skintype
  Arms: Protection Routine 1; Protection Routine 1+2
Behavioral: Experimental: Protection Routine 2 — The sunscreen application instruction is based on a recently developed thorough application instructions for use of sunscreen to counter the problems and deficits of current sunscreen use. It describes every part of the body, the needed volume for that part and application patterns. The package will also include a hat specifically designed for protection and comfort and the availability of a hat will function to increase the use of hat. The hat is simple bucket hat version with a brim, cheap, in light fabric and foldable for easy packing.
  Other Names: Thorough sunscreen and availability of hat
  Arms: Protection Routine 1+2; Protection Routine 2

SUMMARY:
The aim of the study is to test a series of developed effective interventions targeting Danes going on vacation to sunny destinations to decrease sunburn by increasing use of shade, hats, protective clothing, and sunscreen to prevent skin cancer in the Danish population. It has been estimated that up to 90 % of all skin cancers could be avoided by behavioral changes. One of the main sources of UVR exposure in the Danish population is vacations to destinations with high UV index (UVI).

DETAILED DESCRIPTION:
The aim of the study is to test a series of developed effective interventions targeting Danes going on vacation to sunny destinations to decrease sunburn by increasing use of shade, hats, protective clothing, and sunscreen to prevent skin cancer in the Danish population. To achieve the aim of this study we will conduct a randomized controlled trial with four arms during May-Dec 2018. Participants will be Danish adults traveling on vacation in 2018 for a period of 1-3 weeks, recruited from the civil registration system. After enrollment and pretesting, participants will be randomly assigned to one of four experimental conditions. Three experimental groups will receive innovative intervention strategies for promoting sun protection practices during vacation - Protection Routine (1), Protection Routine (2) or both Protection Routine (1+2). The fourth experimental condition will be a minimal treatment control group. The primary outcomes of the trial will be a reduction in frequency of sunburn by adherence to the current sun protection advice from the Danish Cancer Society, i.e., use of shade, hats, protective clothing, and sunscreen as secondary outcomes. We hypothesize that the following two interventions will be able to reduce significantly the UVR exposure and risk of sunburns in Danes going on vacation to destinations with high UVI.

The participants of the study are recruited from the Danish civil registration based system. The study population will represent all groups of the Danish population. Eligibility criteria for the project are persons living in Denmark going on vacation in May-December 2018 and having a smartphone compatible with either apple iOS (version 7.0 or newer) or Google Android (version 4.0 or newer). The period May to December is chosen as it includes all types of vacationers. The summer vacation constitutes the majority of the sunny vacations of the Danes. The period includes both the summer, where Danes typically travel to the Mediterranean area and the winter period where travel patterns change a bit to more exotic areas like Thailand, Egypt and the Canarias Islands. Exclusion criteria are persons younger than 18 years of age.

Sun protective behavior, exposure to UVR and sunburn will be evaluated by use of a questionnaire validated by personal electronic UV-measurements. This newly developed survey tool has made it possible in this project to evaluate the skin cancer interventions, without tracking of development of skin cancer which can take several years to develop after excessive UVR exposure. The short time period from intervention to evaluation minimizes recall bias.

The primary success criteria of the effectiveness of the interventions is a 10 % decrease in sunburn fraction in the intervention groups as compared to the control group in the post-intervention measurement, as shown possible in the pilot study.

Furthermore, we aim to reach completion and response rates of 90 % of the total sample

Secondary success criteria are increased awareness on the risk of skin cancer, increased use of protection (shade, clothes, hat and sunscreen) and decreased outdoor exposure when the UVI is highest between 12 and 3 pm. For all secondary success criteria, we aim for an improvement of 10 % between interventions and control group.

ELIGIBILITY:
Inclusion Criteria:

* Travel for a vacation to a location with higher UVI than Denmark in the trial period (May-December 2018)
* Access to a smartphone compatible with either iOS (version 7 or newer) or Google Android ( version 4.0 or newer)

Exclusion Criteria:

* Physically or mentally uncapable to complete the planned intervention routines

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1548 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Sunburn | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  Any erythema (selfdetermined by questionnaire which is sent within a week after travelling home)

SECONDARY OUTCOMES:
Awareness of skin cancer risk | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  determined by questionnaire which is sent within a week after travelling home
Use of sunprotection;shade | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  determined by questionnaire which is sent within a week after travelling home
Use of sunprotection;clothes | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
Use of sunprotection;hat | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  determined by questionnaire which is sent within a week after travelling home
Use of sunprotection;sunscreen | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  determined by questionnaire which is sent within a week after travelling home
Sunburn body site | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  determined by questionnaire which is sent within a week after travelling home; relation between relevance of sunprotection and sunburned area
Exposure in UV peak hours | Experienced during participants vacationperiod (1-3 weeks within may-dec 2018)
  determined by questionnaire which is sent within a week after travelling home

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Cancer Society, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT03607578/Prot_SAP_000.pdf